CLINICAL TRIAL: NCT03507777
Title: OPtical Coherence Tomography (OCT) Guided Coronary Stent IMplantation Compared to Angiography: a Multicenter Randomized TriaL in PCI
Brief Title: ILUMIEN IV: OPTIMAL Percutaneous Coronary Intervention (PCI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABT-CIP-10233; SJM-CIP-10218 (Other: Abbott Laboratories)
Record Dates: First submitted 2018-04-03; First posted 2018-04-25 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease; Coronary Stenosis; Atherosclerosis; STEMI; STEMI - ST Elevation Myocardial Infarction; NSTEMI - Non-ST Segment Elevation Myocardial Infarction (MI)
Keywords: ABT-CIP-10233; ILUMIEN OPTIS OCT Imaging System; Dragonfly; Optical Coherence Tomography (OCT); Coronary Stent IMplantation; Angiography
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Atherosclerosis; ST Elevation Myocardial Infarction | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Coronary PCI guided by OCT (Active Comparator): Intervention = Coronary stenting with planned drug eluting stent (DES).
  Stenting will be performed with OCT guidance according to the algorithm described in the protocol. OCT imaging is required pre and post stent implantation.
  At the end of the procedure, a final OCT imaging run must be performed.
  Interventions: Device: Coronary PCI guided by OCT
- Coronary PCI guided by Angiography (Active Comparator): Intervention = Coronary stenting with planned drug eluting stent (DES).
  Stenting will be performed with angiography guidance according to local standard practice.
  At the end of the procedure, a blinded OCT shall be performed to document final stent dimensions and results.
  Interventions: Device: Coronary PCI guided by Angiography

INTERVENTIONS:
Device: Coronary PCI guided by OCT — Stent implantation in high-risk or complex lesions in patients with coronary artery disease using OCT guidance
  Other Names: Optical Coherence Tomography
  Arms: Coronary PCI guided by OCT
Device: Coronary PCI guided by Angiography — Stent implantation in high-risk or complex lesions in patients with coronary artery disease using angiography guidance
  Arms: Coronary PCI guided by Angiography

SUMMARY:
The objective of this prospective, single-blind clinical investigation is to demonstrate the superiority of an Optical Coherence Tomography (OCT)-guided stent implantation strategy as compared to an angiography-guided stent implantation strategy in achieving larger post-PCI lumen dimensions and improving clinical cardiovascular outcomes in patients with high-risk clinical characteristics and/or with high-risk angiographic lesions.

ELIGIBILITY:
Inclusion Criteria (all must be present)

1. Subject must be at least 18 years of age.
2. Subject must have evidence of myocardial ischemia (e.g., stable angina, silent ischemia (ischemia in the absence of chest pain or other anginal equivalents), unstable angina, or acute myocardial infarction) suitable for elective PCI.
3. Patients undergoing planned XIENCE stent implantation during a clinically indicated PCI procedure meeting one or more of the following criteria:

   A) High clinical-risk, defined as;

   i. Medication-treated diabetes mellitus, AND/OR

   B) High angiographic-risk lesion(s), with at least one target lesion in each target vessel planned for randomization meeting at least one of the following criteria;

   i. Target lesion is the culprit lesion responsible for either:
   * NSTEMI, defined as a clinical syndrome consistent with an acute coronary syndrome and a minimum troponin of 1 ng/dL (may or may not have returned to normal), OR
   * STEMI >24 hours from the onset of ischemic symptoms

   ii. long or multiple lesions (defined as intended total stent length in any single target vessel ≥28 mm),

   Note: For a long target lesion, this would permit treatment by a single long stent or overlapping stents.

   Note: For up to two target lesions located in a single target vessel and treated with non-overlapping stents, they may be located in a continuous vessel or split up between a main vessel and a side branch.

   iii. bifurcation intended to be treated with 2 planned stents (i.e. in both the main branch and side branch), and where the planned side branch stent is ≥ 2.5 mm in diameter by angiographic visual estimation.

   iv. angiographic severe calcification (defined as angiographically visible calcification on both sides of the vessel wall in the absence of cardiac motion),

   v. chronic total occlusion (CTO) (enrolment and randomization in this case performed only after successful antegrade wire escalation crossing and pre-dilatation)

   vi. in-stent restenosis of diffuse or multi-focal pattern. Lesion must be at or within the existing stent margin(s) and have angiographically visually-assessed DS ≥70% or DS ≥50% with non-invasive or invasive evidence of ischemia
4. All target lesions (those lesions to be randomized) must have a visually estimated or quantitatively assessed %DS of either ≥70%, or ≥50% plus one or more of the following: an abnormal functional test (e.g. fractional flow reserve, stress test) signifying ischemia in the distribution of the target lesion(s) or biomarker positive ACS with plaque disruption or thrombus.

   Note: For purposes of study eligibility, a minimum troponin of 1 ng/dL at the time of screening will be considered biomarker positive.
5. All target lesions must be planned for treatment with only ≥2.5 mm and ≤3.5 mm stents and post-dilatation balloons based on pre-PCI angiographic visual estimation.
6. No more than 2 target lesions requiring PCI are present in any single vessel., and no more than 2 target vessels are allowed. Thus, up to 4 randomized target lesions per patient in a maximum of 2 target vessels are allowed, including branches. The intended target lesions will be declared just prior to randomization.

   Note: A lesion is defined as any segment(s) of the coronary tree, no matter how long, which is planned to be covered with one contiguous length of stent, whether single or overlapped. A bifurcation counts as a single lesion even if the side branch is planned to be treated.

   Note: All lesions in a randomized target vessel that are intended to be treated by PCI are designated as target lesions, and at least one target lesion in each randomized target vessel must meet angiographic high-risk inclusion criteria summarized above in 3B). The only exception is for patients who qualify for the trial on the basis of medication-treated diabetes, in which case no target lesion is required to meet angiographic high-risk inclusion criteria.
7. All target lesions intended to be treated by PCI in the target vessel are amenable to OCT-guided PCI.

   Example: If a qualifying angiographic high-risk lesion is in the proximal LAD, and there is a second target lesion in the distal LAD which is a focal lesion not otherwise meeting high-risk criteria, both the proximal LAD and distal LAD lesions must be amenable to OCT (e.g. no excessive tortuosity or calcification precluding delivering the OCT catheter), and each lesion must undergo OCT-guided stenting. Otherwise the vessel should be excluded from randomization.
8. Subject must provide written Informed Consent prior to any study related procedure.

Exclusion Criteria (none may be present)

Clinical exclusion criteria:

1. STEMI ≤24 hours from the onset of ischemic symptoms
2. Creatinine clearance ≤30 ml/min/1.73 m^2 (as calculated by MDRD formula for estimated GFR) and not on dialysis. Note: chronic dialysis dependent patients are eligible for enrolment regardless of creatinine clearance.
3. Hypotension, shock or need for mechanical support or intravenous vasopressors at the time the patient would be undergoing the index procedure.
4. CHF (Killip class ≥2 or NYHA class ≥3)
5. LVEF ≤30% by the most recent imaging test within 3 months prior to procedure. If no LVEF test result within 3 months is available, it must be assessed by echocardiography, multiple gated acquisition (MUGA), magnetic resonance imaging (MRI), ventriculography (LV gram) or other method.
6. Unstable ventricular arrhythmias
7. Inability to take DAPT (both aspirin and a P2Y12 inhibitor) for at least 12 months in the patient presenting with an ACS, or at least 6 months in the patient presenting with stable CAD, unless the patient is also taking chronic oral anticoagulation in which case a shorter duration of DAPT may be prescribed per local standard of care.
8. Planned major cardiac or non-cardiac surgery within 24 months after the index procedure.

   Note: Major surgery is any invasive operative procedure in which an extensive resection is performed, e.g. a body cavity is entered, organs are removed, or normal anatomy is altered.

   Note: Minor surgery is an operation on the superficial structures of the body or a manipulative procedure that does not involve a serious risk. Planned minor surgery is not excluded.
9. Prior PCI within the target vessel within 12 months

   Note: Prior PCI within the target vessel within 12 months is allowed for in-stent restenosis (target lesion is the prior PCI site) if no more than one layer of previously implanted stent is present.

   Note: In-stent restenosis involving two or more layers of stent implanted at any time prior to index procedure (i.e. an earlier episode of in-stent restenosis previously treated with a second stent) is excluded.
10. Any planned PCI within the target vessel(s) within 24 months after the study procedure, other than a planned staged intervention in a second randomized target vessel.

    Note: Planned staged interventions must be noted at the time of randomization, and the decision to stage may be modified within 24 hours of completion of the index PCI.

    Note: PCI in non-target vessels is permitted >48 hours after the index procedure.
11. Any prior PCI in a non-target vessel within 24 hours before the study procedure, or within previous 30 days if unsuccessful or complicated.

    Note: Patients requiring non-target vessel PCI may be enrolled and the non-target vessel(s) may be treated in the same index procedure as the randomized lesions (in all cases prior to randomization), as long as treatment of the lesion(s) in the non-target vessel is successful and uncomplicated.

    Successful and uncomplicated definition for non-target vessel treatment during the index procedure: Angiographic diameter stenosis <10% for all treated non-target lesions, with TIMI III flow in this vessel, without final dissection ≥ NHLBI type B, perforation anytime during the procedure, prolonged chest pain (>5 minutes) or prolonged ST-segment elevation or depression (>5 minutes), or cardiac arrest or need for defibrillation or cardioversion or hypotension/heart failure requiring mechanical or intravenous hemodynamic support or intubation).
12. Subject has known hypersensitivity or contraindication to any of the study drugs (including all P2Y12 inhibitors, one or more components of the study devices, including everolimus, cobalt, chromium, nickel, platinum, tungsten, acrylic and fluoropolymers, or radiocontrast dye) that cannot be adequately pre-medicated.
13. Subject has received a solid organ transplant which is functioning or is active on a waiting list for any solid organ transplants with expected transplantation within 24 months.
14. Subject is receiving immunosuppressant therapy or has known immunosuppressive or severe autoimmune disease that requires chronic immunosuppressive therapy (e.g., human immunodeficiency virus, systemic lupus erythematosus, etc.). Note: corticosteroids are not included as immunosuppressant therapy.
15. Subject has previously received or is scheduled to receive radiotherapy to a coronary artery (vascular brachytherapy), or the chest/mediastinum.
16. Subject has a platelet count <100,000 cells/mm^3 or >700,000 cells/mm^3.
17. Subject has a documented or suspected hepatic disorder as defined as cirrhosis or Child-Pugh ≥ Class B.
18. Subject has a history of bleeding diathesis or coagulopathy, or has had a significant gastro-intestinal or significant urinary bleed within the past six months.
19. Subject has had a cerebrovascular accident or transient ischemic neurological attack (TIA) within the past six months, or any prior intracranial bleed, or any permanent neurologic defect, or any known intracranial pathology (e.g., aneurysm, arteriovenous malformation, etc.).
20. Subject has extensive peripheral vascular disease that precludes safe 6 French sheath insertion. Note: femoral arterial disease does not exclude the patient if radial access may be used.
21. Subject has life expectancy <2 years for any non-cardiac cause.
22. Subject is currently participating in another investigational drug or device clinical study that has not yet completed its primary endpoint.
23. Pregnant or nursing subjects and those who plan pregnancy in the period up to 2 years following index procedure. Female subjects of child-bearing potential must have a negative pregnancy test done within 7 days prior to the index procedure per site standard test.
24. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.

Angiographic exclusion criteria

1. Syntax score ≥33, unless a formal meeting of the Heart Team, including a cardiac surgeon, concludes that PCI is appropriate.
2. Planned use of any stent <2.5 mm in a target vessel based on visual estimation (note: a smaller stent may be used in a bail-out scenario - e.g. to treat a distal dissection - but its use cannot be planned prior to enrolment)
3. Planned use of a stent or post-dilatation balloon ≥3.75 mm for the target lesion
4. Severe vessel tortuosity or calcification in a target vessel such that it is unlikely that the OCT catheter can be delivered (note: severe vessel calcification is allowed if it is expected that the OCT catheter can be delivered at baseline or after vessel preparation with balloon pre-dilatation or atherectomy)
5. The target vessel has a lesion with DS ≥ 50% that is not planned for treatment at the time of index procedure.
6. The target lesion is in the left main coronary artery
7. The target lesion is in a bypass graft conduit. Note: A native coronary artery may be randomized if a prior bypass graft conduit to the vessel is totally occluded, but not if it is patent.
8. The target lesion is an ostial RCA stenosis
9. The target lesion is a stent thrombosis
10. Planned use of any stent other than Xience in a target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2487 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregg W Stone, MD, Study Chair — Icahn School of Medicine at Mount Sinai; Ulf Landmesser, MD, Principal Investigator — Charite University, Berlin, Germany; Ziad A Ali, MD, DPhil, Principal Investigator — St Francis Hospital and Heart Center
Locations (90):
- United States (42):
  - University Hospital - Univ. of Alabama at Birmingham (UAB), Birmingham, Alabama
  - Scottsdale Healthcare Shea, Scottsdale, Arizona
  - Mills-Peninsula Medical Center, Burlingame, California
  - John Muir Medical Center, Concord, California
  - Scripps Health, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California - Davis Medical Center, Sacramento, California
  - University of California at San Diego (UCSD) Medical Center, San Diego, California
  - Stanford University Medical Center, Stanford, California
  - The Cardiac & Vascular Institute Research Foundation, LLC, Gainesville, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Kansas University Medical Center, Kansas City, Kansas
  - Via Christi Regional Medical Center - St. Francis Campus, Wichita, Kansas
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Massachusetts Medical Center, Worcester, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - St. Patrick Hospital, Missoula, Montana
  - Buffalo General Hospital, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - New York Presbyterian Hospital/Columbia University, New York, New York
  - St. Francis Hospital, Roslyn, New York
  - Montefiore Medical Center - Moses Division, The Bronx, New York
  - Mission Health & Hospitals, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Eastern Cardiology, Greenville, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - St. Charles Medical Center, Bend, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Centennial Heart Cardiovascular Consultants, Nashville, Tennessee
  - Austin Heart, Austin, Texas
  - Memorial Hermann Hospital, Houston, Texas
  - McKay-Dee Heart Services, Ogden, Utah
  - Providence Everett Medical Center, Everett, Washington
  - Swedish Medical Center, Seattle, Washington
- Australia (3):
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Eastern Heart Clinic - Prince of Wales Hospital, Randwick
- Belgium (2):
  - Onze-Lieve-Vrouwziekenhuis Campus Aalst, Aalst, Eflndrs
  - UZ Gasthuisberg, Leuven, Flemish Brabant
- Canada (6):
  - Royal Jubilee Hospital, Victoria, British Columbia
  - QE II Health Sciences, Halifax, Nova Scotia
  - Hamilton Health Science Centre, Hamilton, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - CHUM, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
- Skejby University Hospital, Aarhus, Denmark
- France (3):
  - Hopital Cardiovasculaire et Pneumologique Louis Pradel, Lyon, Auvergne-Rhône-Alpes
  - CHU Gabriel Montpied, Clermont-Ferrand, Auvergn
  - CHU de Besancon - Jean Minjoz, Besançon, Franche-Comte
- Germany (5):
  - Kliniken der Friedrich-Alexander-Universitat, Erlangen, Bavaria
  - Deutsches Herzzentrum München des Freistaates Bayern, Munich, Bavaria
  - Klinikum der Justus-Liebig-Universität, Giessen, Hesse
  - UNIVERSITATSMEDIZIN der Johannes Gutenberg-Universität Mainz, Mainz, Rhinela
  - Universitätsmedizin Berlin - Campus Benjamin Franklin (CBF), Berlin
- Hong Kong (3):
  - Prince of Wales Hospital, Hong Kong, HK SAR
  - Queen Elizabeth Hospital, Hong Kong, HK SAR
  - Queen Mary Hospital, Hong Kong, HK SAR
- India (4):
  - Apollo Hospital, Chennai, Tamil Nadu
  - The Madras Medical Mission, Chennai, Tamil Nadu
  - Postgraduate Institute of Medical Education & Research, Chandigarh
  - Max Super Specialty Hospital, New Delhi
- Italy (4):
  - Policlinico Universitario A. Gemelli, Rome, Lazio
  - Az. Osp. S. Giovanni Addolorata, Rome, Lazio
  - Ospedale Papa Giovanni XXIII, Bergamo, Lombard
  - Centro Cardiologico Monzino, Milan, Lombard
- Wakayama Medical University, Wakayama, Japan
- Netherlands (2):
  - Albert Schweitzer Ziekenhuis, Dordrecht, South Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland
- New Zealand (2):
  - Christchurch Hospital, Christchurch, Canterbury
  - Wellington Hospital, Wellington
- Hospital Santa Marta, Lisbon, Lisbon District, Portugal
- National University Hospital, Singapore, Central, Singapore
- Spain (2):
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario de la Princesa, Madrid
- Sahlgrenska University Hospital - Gothenburg, Gothenburg, Vastra, Sweden
- Switzerland (2):
  - Center Inselspital Bern, Bern
  - Luzerner Kantonsspital, Lucerne
- Taiwan (2):
  - National Taiwan University Hospital, Taipei, Ntaiwan
  - Taipei Veterans General Hospital (VGH), Taipei, Ntaiwan
- United Kingdom (3):
  - Bristol Royal Infirmary, Bristol, West Midland
  - Papworth Hospital NHS Foundation Trust, Cambridge
  - Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Johnson TW, Bergmark BA, Croce K, Pellegrini D, Maehara A, Gori T, Pinilla-Echeverri N, Wollmuth J, Gonzalo N, Kao HL, Guagliumi G, Phalakornkule K, Ediebah D, McNutt J, Chiu WC, Op den Buijs J, Buccola J, Landmesser U, Ali Z, Stone GW, Jeremias A. Impact of Optical Coherence Tomography-Based Post-PCI Physiology Assessment to Predict Clinical Outcomes: An ILUMIEN-IV Substudy. J Am Coll Cardiol. 2025 Jul 15;86(2):93-102. doi: 10.1016/j.jacc.2025.05.019. Epub 2025 May 22. PMID 40406943
- [Derived] Ali ZA, Landmesser U, Maehara A, Shin D, Sakai K, Matsumura M, Shlofmitz RA, Calligaris G, Maksoud A, Abdelwahed YS, Canova P, Gonzalo N, Alfonso F, Fall KN, Chehab B, McGreevy RJ, McNutt RW, Nie H, Wang J, Buccola J, Stone GW; ILUMIEN IV Investigators. Safety and Efficacy of Cobalt Chromium Everolimus-Eluting Stents for Treatment of In-Stent Restenosis: An ILUMIEN IV Substudy. J Am Heart Assoc. 2025 Jun 3;14(11):e039482. doi: 10.1161/JAHA.124.039482. Epub 2025 May 22. PMID 40401609
- [Derived] Ali ZA, Landmesser U, Maehara A, Shin D, Sakai K, Matsumura M, Shlofmitz RA, Leistner D, Canova P, Alfonso F, Fabbiocchi F, Guagliumi G, Price MJ, Hill JM, Akasaka T, Prati F, Bezerra HG, Wijns W, McGreevy RJ, McNutt RW, Nie H, Phalakornkule K, Buccola J, Stone GW; ILUMIEN IV Investigators. OCT-Guided vs Angiography-Guided Coronary Stent Implantation in Complex Lesions: An ILUMIEN IV Substudy. J Am Coll Cardiol. 2024 Jul 23;84(4):368-378. doi: 10.1016/j.jacc.2024.04.037. Epub 2024 May 15. PMID 38759907
- [Derived] Ali ZA, Landmesser U, Maehara A, Matsumura M, Shlofmitz RA, Guagliumi G, Price MJ, Hill JM, Akasaka T, Prati F, Bezerra HG, Wijns W, Leistner D, Canova P, Alfonso F, Fabbiocchi F, Dogan O, McGreevy RJ, McNutt RW, Nie H, Buccola J, West NEJ, Stone GW; ILUMIEN IV Investigators. Optical Coherence Tomography-Guided versus Angiography-Guided PCI. N Engl J Med. 2023 Oct 19;389(16):1466-1476. doi: 10.1056/NEJMoa2305861. Epub 2023 Aug 27. PMID 37634188
- [Derived] Ali Z, Landmesser U, Karimi Galougahi K, Maehara A, Matsumura M, Shlofmitz RA, Guagliumi G, Price MJ, Hill JM, Akasaka T, Prati F, Bezerra HG, Wijns W, Mintz GS, Ben-Yehuda O, McGreevy RJ, Zhang Z, Rapoza RR, West NEJ, Stone GW. Optical coherence tomography-guided coronary stent implantation compared to angiography: a multicentre randomised trial in PCI - design and rationale of ILUMIEN IV: OPTIMAL PCI. EuroIntervention. 2021 Jan 20;16(13):1092-1099. doi: 10.4244/EIJ-D-20-00501. PMID 32863246

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first randomized subject was enrolled in the study on May 17, 2018. The trial completed enrollment on December 29, 2020 with a total of 2487 randomized subjects. The randomized subjects, who were enrolled at 80 sites in 18 countries, were comprised of 1233 subjects assigned to the OCT-guided PCI arm and 1254 subjects in the angiography-guided PCI arm.
Pre-assignment Details: In this study, the total number of randomized participants were 2487, out of which 1233 were assigned to OCT guidance and 1254 were assigned to angiography guidance.
Groups:
- Coronary PCI Guided by OCT: Intervention = Coronary stenting with planned drug eluting stent (DES).
  Stenting will be performed with OCT guidance according to the algorithm described in the protocol. OCT imaging is required pre and post stent implantation.
  At the end of the procedure, a final OCT imaging run must be performed.
  Coronary PCI guided by OCT: Stent implantation in high-risk or complex lesions in patients with coronary artery disease using OCT guidance
- Coronary PCI Guided by Angiography: Intervention = Coronary stenting with planned drug eluting stent (DES).
  Stenting will be performed with angiography guidance according to local standard practice.
  At the end of the procedure, a blinded OCT shall be performed to document final stent dimensions and results.
  Coronary PCI guided by Angiography: Stent implantation in high-risk or complex lesions in patients with coronary artery disease using angiography guidance
Period: Overall Study
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by Angiography
Started | 1233 | 1254
Completed | 1189 | 1184
Not Completed | 44 | 70
Not completed — Lost to Follow-up | 5 | 7
Not completed — Withdrawal by Subject | 6 | 11
Not completed — Death | 30 | 44
Not completed — Other Reasons | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by Angiography | Total
Number analyzed (Participants) | 1233 | 1254 | 2487
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.5 (10.5) | 65.7 (10.3) | 65.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 265 | 298 | 563
  Male | 968 | 956 | 1924
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 61 | 67 | 128
  Not Hispanic or Latino | 870 | 867 | 1737
  Unknown or Not Reported | 302 | 320 | 622
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 271 participants in the OCT arm and 298 participants in the angio arm declined to specify Race or the data were not released due to local regulations.
  Participants
    American Indian or Alaska Native | 3 | 4 | 7
    Asian | 152 | 156 | 308
    Native Hawaiian or Other Pacific Islander | 6 | 6 | 12
    Black or African American | 42 | 43 | 85
    White | 759 | 744 | 1503
    More than one race | 0 | 3 | 3
    Unknown or Not Reported | 271 | 298 | 569
Region of Enrollment [Number; unit: participants]
  United States | 451 | 458 | 909
  Canada | 53 | 55 | 108
  Europe | 540 | 553 | 1093
  Pacifica | 189 | 188 | 377
Hypertension req. Medication [Number; unit: participants] | 880 | 928 | 1808

OUTCOME MEASURES:

1. Primary Outcome: Imaging Outcome (Powered): Minimal Stent Area (MSA)
Description: Minimal Stent Area (per target lesion basis) assessed by OCT in each randomized arm, measured at an independent OCT core laboratory blinded to imaging modality assignment.
Time Frame: Final Post-PCI Measurement (average of 24 hours).
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: lesions
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 1147 | 1201
Number analyzed (lesions) | 1147 | 1201
mm^2 | 5.72 (2.04) | 5.36 (1.87)
Statistical Analysis 1: Comparison: Coronary PCI Guided by OCT vs Coronary PCI Guided by Angiography; Test type: Superiority; p < 0.0001, Linear mixed model

2. Primary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: Time-to-first event rate of the composite outcome of cardiac death, target vessel myocardial infarction (TV-MI), or ischemia-driven target vessel revascularization (ID-TVR), will be assessed.
Time Frame: At 2 years
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: participants who experienced the event
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 1233 | 1254
participants who experienced the event | 88 | 99
Statistical Analysis 1: Comparison: Coronary PCI Guided by OCT vs Coronary PCI Guided by Angiography; Test type: Superiority; p = 0.2487, A Cox regression model

3. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF) Excluding Periprocedural MI (Powered)
Description: Time-to-first event rate of composite outcome of cardiac death, target vessel-related spontaneous myocardial infarction, or ischemia-driven target vessel revascularization (ID-TVR) will be assessed.
Time Frame: At 2 years
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: participants who experienced the event
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 1233 | 1254
participants who experienced the event | 74 | 82
Statistical Analysis 1: Comparison: Coronary PCI Guided by OCT vs Coronary PCI Guided by Angiography; Test type: Superiority; p = 0.2952, A Cox regression model

4. Secondary Outcome: The Results of Adjudicated Clinical Outcomes to 2 Years in the Randomized Population
Description: The results of adjudicated clinical outcomes to 2 years in the randomized population by Kaplan-Meier assessment.
Time Frame: 2 years
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 1233 | 1254
participants
  All Death | 32 | 44
  All MI | 57 | 72
  All Revascularization | 112 | 120
  All Death, All MI, All Revascularization (DMR) | 171 | 187
  TVF | 88 | 99
  TVF excluding PPMI | 74 | 82
  TLF | 76 | 86

5. Secondary Outcome: The Number of Participants With Stent Thrombosis
Description: The results of adjudicated clinical outcomes to 2 years in the randomized population by Kaplan-Meier assessment.
Time Frame: 2 years
Population: The number of participants analyzed includes subjects who were available at that time of analysis
Measure: Number; unit: participants
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by Angiography
Number analyzed (Participants) | 1233 | 1254
participants
  Definite | 5 | 14
  Definite/Probable | 6 | 17

ADVERSE EVENTS:
Time Frame: 2 years
Description: There are 8 pre-specified categories of site-reported AE (dissection, hypotension, myocardial infarction, stent thrombosis, stroke, target lesion revascularization (TLR), TVR and vessel perforation) and a broad category designated as "Other". AEs falling into the "Other" category are categorized to standard medical terms using the Medical Dictionary for Regulatory Activities (MedDRA) code and preferred term.
Arm/Group | Coronary PCI Guided by OCT | Coronary PCI Guided by Angiography
All-Cause Mortality (participants affected / at risk) | 33/1233 | 44/1254
Serious Adverse Events (participants affected / at risk) | 405/1233 | 411/1254
Other Adverse Events (participants affected / at risk) | 71/1233 | 73/1254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Coronary PCI Guided by OCT (N=1233) | Coronary PCI Guided by Angiography (N=1254)
ANAEMIA (Blood and lymphatic system disorders) | 12 | 6
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 3 | 0
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 2 | 6
ANGINA PECTORIS (Cardiac disorders) | 25 | 17
ANGINA UNSTABLE (Cardiac disorders) | 21 | 23
AORTIC VALVE STENOSIS (Cardiac disorders) | 1 | 3
ARRHYTHMIA (Cardiac disorders) | 2 | 1
ARTERIOSCLEROSIS CORONARY ARTERY (Cardiac disorders) | 2 | 1
ARTERIOSPASM CORONARY (Cardiac disorders) | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 13 | 16
ATRIAL FLUTTER (Cardiac disorders) | 4 | 1
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 2 | 3
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 1
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 0 | 1
BRADYCARDIA (Cardiac disorders) | 6 | 3
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 0 | 1
CARDIAC ARREST (Cardiac disorders) | 3 | 1
CARDIAC FAILURE (Cardiac disorders) | 7 | 6
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 2
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 2 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 3 | 3
CARDIAC TAMPONADE (Cardiac disorders) | 1 | 0
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 1 | 0
CARDIOMYOPATHY (Cardiac disorders) | 0 | 2
CARDIORENAL SYNDROME (Cardiac disorders) | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 12 | 8
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 2 | 2
CORONARY ARTERY STENOSIS (Cardiac disorders) | 5 | 5
CORONARY NO-REFLOW PHENOMENON (Cardiac disorders) | 1 | 0
DRESSLER'S SYNDROME (Cardiac disorders) | 1 | 0
EXTRASYSTOLES (Cardiac disorders) | 0 | 2
INTRACARDIAC THROMBUS (Cardiac disorders) | 0 | 1
ISCHAEMIC CARDIOMYOPATHY (Cardiac disorders) | 1 | 1
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 1
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 1 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 26 | 43
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 2 | 5
PALPITATIONS (Cardiac disorders) | 5 | 4
PERICARDIAL EFFUSION (Cardiac disorders) | 2 | 2
PERICARDITIS (Cardiac disorders) | 0 | 1
PULSELESS ELECTRICAL ACTIVITY (Cardiac disorders) | 1 | 1
SICK SINUS SYNDROME (Cardiac disorders) | 2 | 3
SINUS ARREST (Cardiac disorders) | 1 | 1
SINUS TACHYCARDIA (Cardiac disorders) | 1 | 0
STRESS CARDIOMYOPATHY (Cardiac disorders) | 1 | 0
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 1
VENTRICULAR FIBRILLATION (Cardiac disorders) | 4 | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 1 | 4
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 0 | 1
HYDROCELE (Congenital, familial and genetic disorders) | 0 | 1
MUSCULAR DYSTROPHY (Congenital, familial and genetic disorders) | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 0 | 1
HYPERPARATHYROIDISM (Endocrine disorders) | 0 | 1
INAPPROPRIATE ANTIDIURETIC HORMONE SECRETION (Endocrine disorders) | 0 | 1
CATARACT (Eye disorders) | 3 | 3
DIABETIC RETINOPATHY (Eye disorders) | 0 | 1
DIPLOPIA (Eye disorders) | 0 | 1
EYE PAIN (Eye disorders) | 1 | 0
GLAUCOMA (Eye disorders) | 0 | 1
HYPHAEMA (Eye disorders) | 0 | 1
RETINAL VEIN OCCLUSION (Eye disorders) | 0 | 1
VISION BLURRED (Eye disorders) | 1 | 0
VISUAL ACUITY REDUCED (Eye disorders) | 0 | 1
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 11 | 3
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 4
ASCITES (Gastrointestinal disorders) | 1 | 0
COLITIS (Gastrointestinal disorders) | 0 | 1
DUODENITIS (Gastrointestinal disorders) | 1 | 0
ENTEROCOLITIS HAEMORRHAGIC (Gastrointestinal disorders) | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 2 | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 10 | 11
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0
HIATUS HERNIA (Gastrointestinal disorders) | 0 | 1
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 1
INTESTINAL ISCHAEMIA (Gastrointestinal disorders) | 1 | 0
INTESTINAL POLYP (Gastrointestinal disorders) | 0 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 2
MELAENA (Gastrointestinal disorders) | 1 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1
ODYNOPHAGIA (Gastrointestinal disorders) | 1 | 0
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 1
PANCREATIC FISTULA (Gastrointestinal disorders) | 1 | 0
PANCREATIC MASS (Gastrointestinal disorders) | 1 | 0
PANCREATITIS (Gastrointestinal disorders) | 0 | 2
PANCREATITIS ACUTE (Gastrointestinal disorders) | 1 | 1
PERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 4 | 0
RECTAL POLYP (Gastrointestinal disorders) | 1 | 1
RETROPERITONEAL HAEMATOMA (Gastrointestinal disorders) | 0 | 1
RETROPERITONEAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
UMBILICAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 | 1
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3 | 1
ASTHENIA (General disorders) | 0 | 3
CATHETER SITE HAEMORRHAGE (General disorders) | 1 | 0
CHEST DISCOMFORT (General disorders) | 8 | 2
CHEST PAIN (General disorders) | 75 | 50
DEATH (General disorders) | 9 | 17
GAIT DISTURBANCE (General disorders) | 0 | 1
HERNIA (General disorders) | 0 | 1
IMPAIRED HEALING (General disorders) | 0 | 1
MALAISE (General disorders) | 1 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 3 | 4
PYREXIA (General disorders) | 5 | 5
THROMBOSIS IN DEVICE (General disorders) | 6 | 9
VESSEL PUNCTURE SITE HAEMORRHAGE (General disorders) | 1 | 0
BILE DUCT OBSTRUCTION (Hepatobiliary disorders) | 0 | 1
CHOLANGITIS (Hepatobiliary disorders) | 1 | 2
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 3
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 1
HEPATITIS ACUTE (Hepatobiliary disorders) | 1 | 0
ANAPHYLACTIC REACTION (Immune system disorders) | 1 | 0
TRANSPLANT REJECTION (Immune system disorders) | 0 | 1
ABSCESS LIMB (Infections and infestations) | 0 | 1
ANAL ABSCESS (Infections and infestations) | 1 | 0
APPENDICITIS (Infections and infestations) | 1 | 1
BACTERAEMIA (Infections and infestations) | 1 | 0
CELLULITIS (Infections and infestations) | 1 | 4
CLOSTRIDIAL INFECTION (Infections and infestations) | 1 | 0
CORONA VIRUS INFECTION (Infections and infestations) | 15 | 18
CYSTITIS (Infections and infestations) | 0 | 2
DIABETIC FOOT INFECTION (Infections and infestations) | 1 | 0
EMPYEMA (Infections and infestations) | 0 | 1
ENDOCARDITIS (Infections and infestations) | 0 | 2
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 | 0
ERYSIPELAS (Infections and infestations) | 1 | 0
FURUNCLE (Infections and infestations) | 0 | 1
GALLBLADDER ABSCESS (Infections and infestations) | 0 | 1
GANGRENE (Infections and infestations) | 2 | 1
GASTROENTERITIS (Infections and infestations) | 2 | 1
HAEMATOMA INFECTION (Infections and infestations) | 0 | 1
HEPATIC CYST INFECTION (Infections and infestations) | 0 | 1
HERPES ZOSTER OPHTHALMIC (Infections and infestations) | 0 | 1
INFECTION (Infections and infestations) | 1 | 4
INFLUENZA (Infections and infestations) | 1 | 0
LOBAR PNEUMONIA (Infections and infestations) | 0 | 1
LOCALISED INFECTION (Infections and infestations) | 0 | 2
OSTEOMYELITIS (Infections and infestations) | 1 | 2
PERITONITIS (Infections and infestations) | 1 | 0
PHARYNGITIS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 16 | 6
PNEUMONIA PRIMARY ATYPICAL (Infections and infestations) | 0 | 1
PULMONARY SEPSIS (Infections and infestations) | 0 | 1
PYELONEPHRITIS (Infections and infestations) | 1 | 0
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 0 | 1
SEPSIS (Infections and infestations) | 6 | 2
SEPTIC ENCEPHALOPATHY (Infections and infestations) | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 2
SINUSITIS (Infections and infestations) | 2 | 0
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1
TOOTH INFECTION (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 5 | 3
UROSEPSIS (Infections and infestations) | 3 | 2
VESTIBULAR NEURONITIS (Infections and infestations) | 0 | 2
VIRAL INFECTION (Infections and infestations) | 1 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
ARTERIOVENOUS FISTULA THROMBOSIS (Injury, poisoning and procedural complications) | 1 | 1
BACK INJURY (Injury, poisoning and procedural complications) | 0 | 1
CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 2 | 0
FALL (Injury, poisoning and procedural complications) | 8 | 8
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
HEAD INJURY (Injury, poisoning and procedural complications) | 2 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 | 2
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 4 | 6
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 | 1
LACERATION (Injury, poisoning and procedural complications) | 1 | 0
PLAQUE SHIFT (Injury, poisoning and procedural complications) | 1 | 0
POST PROCEDURAL HAEMATURIA (Injury, poisoning and procedural complications) | 0 | 1
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0
SKIN WOUND (Injury, poisoning and procedural complications) | 0 | 1
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 1
SUBDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 1 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 | 1
TONGUE INJURY (Injury, poisoning and procedural complications) | 0 | 1
ULNA FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
URETHRAL INJURY (Injury, poisoning and procedural complications) | 0 | 1
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 4 | 2
BLOOD CREATININE INCREASED (Investigations) | 1 | 1
BLOOD PRESSURE DECREASED (Investigations) | 1 | 0
BLOOD PRESSURE INCREASED (Investigations) | 1 | 0
CARDIAC ENZYMES INCREASED (Investigations) | 3 | 1
CARDIAC STRESS TEST ABNORMAL (Investigations) | 2 | 3
CORONAVIRUS TEST POSITIVE (Investigations) | 1 | 0
EJECTION FRACTION ABNORMAL (Investigations) | 1 | 0
HAEMOGLOBIN ABNORMAL (Investigations) | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 1 | 2
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1 | 1
SINGLE PHOTON EMISSION COMPUTERISED TOMOGRAM ABNORMAL (Investigations) | 0 | 1
TROPONIN INCREASED (Investigations) | 5 | 9
VIRAL TEST (Investigations) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 0
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 | 1
ELECTROLYTE IMBALANCE (Metabolism and nutrition disorders) | 0 | 1
FLUID OVERLOAD (Metabolism and nutrition disorders) | 1 | 1
FOOD INTOLERANCE (Metabolism and nutrition disorders) | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 2
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 | 1
HYPERVOLAEMIA (Metabolism and nutrition disorders) | 2 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 2
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 3
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
BURSITIS (Musculoskeletal and connective tissue disorders) | 1 | 0
COMPARTMENT SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
LUMBAR SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 3 | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 2
MYOPATHY (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 3 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3 | 2
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 1 | 1
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
PSEUDARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 2
PUBIC PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
SPINAL COLUMN STENOSIS (Musculoskeletal and connective tissue disorders) | 1 | 1
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 1 | 0
TENDON DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 1
ADENOCARCINOMA PANCREAS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ADRENAL ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BILIARY NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
GASTRIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LIP AND/OR ORAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
LUNG SQUAMOUS CELL CARCINOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
MALIGNANT NEOPLASM OF RENAL PELVIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MYELODYSPLASTIC SYNDROME (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NASAL CAVITY CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
RECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CAROTID ARTERIOSCLEROSIS (Nervous system disorders) | 0 | 1
CAROTID ARTERY DISEASE (Nervous system disorders) | 1 | 0
CAROTID ARTERY STENOSIS (Nervous system disorders) | 1 | 1
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 9 | 10
COGNITIVE DISORDER (Nervous system disorders) | 1 | 1
CONVULSION (Nervous system disorders) | 0 | 2
DEMENTIA (Nervous system disorders) | 1 | 0
DEMENTIA ALZHEIMER'S TYPE (Nervous system disorders) | 0 | 1
DIZZINESS (Nervous system disorders) | 3 | 3
DYSARTHRIA (Nervous system disorders) | 1 | 0
ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
EPILEPSY (Nervous system disorders) | 0 | 2
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 | 1
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 | 0
HEADACHE (Nervous system disorders) | 0 | 1
HYPOAESTHESIA (Nervous system disorders) | 1 | 1
HYPOXIC-ISCHAEMIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
PARAESTHESIA (Nervous system disorders) | 0 | 1
PARKINSON'S DISEASE (Nervous system disorders) | 0 | 2
PRESYNCOPE (Nervous system disorders) | 0 | 4
RADICULITIS CERVICAL (Nervous system disorders) | 1 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 | 1
SYNCOPE (Nervous system disorders) | 11 | 12
TOXIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 3 | 1
VERTEBRAL ARTERY DISSECTION (Nervous system disorders) | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 1 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 1 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 1 | 0
DYSURIA (Renal and urinary disorders) | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 5 | 2
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 2 | 3
RENAL FAILURE ACUTE (Renal and urinary disorders) | 3 | 3
RENAL FAILURE CHRONIC (Renal and urinary disorders) | 1 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 1
URETHRAL STENOSIS (Renal and urinary disorders) | 0 | 1
URINARY RETENTION (Renal and urinary disorders) | 2 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 2 | 2
UTERINE PROLAPSE (Reproductive system and breast disorders) | 1 | 0
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 | 0
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2 | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 2 | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 26 | 29
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 3 | 3
HYPERCAPNIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 2
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 | 4
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3 | 2
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 2 | 3
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 3
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SYSTEMIC SCLEROSIS PULMONARY (Respiratory, thoracic and mediastinal disorders) | 1 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 2 | 0
AORTIC VALVE REPLACEMENT (Surgical and medical procedures) | 0 | 1
ARTERIAL STENT INSERTION (Surgical and medical procedures) | 0 | 1
CARDIAC PACEMAKER INSERTION (Surgical and medical procedures) | 1 | 0
CORONARY ARTERIAL STENT INSERTION (Surgical and medical procedures) | 0 | 1
CORONARY ARTERY BYPASS (Surgical and medical procedures) | 1 | 2
CORONARY REVASCULARISATION (Surgical and medical procedures) | 14 | 19
DEBRIDEMENT (Surgical and medical procedures) | 0 | 1
FOOT AMPUTATION (Surgical and medical procedures) | 1 | 0
HIP ARTHROPLASTY (Surgical and medical procedures) | 3 | 1
HOSPITALISATION (Surgical and medical procedures) | 0 | 1
KNEE ARTHROPLASTY (Surgical and medical procedures) | 0 | 3
NEPHRECTOMY (Surgical and medical procedures) | 0 | 1
PROSTATECTOMY (Surgical and medical procedures) | 1 | 0
RENAL TRANSPLANT (Surgical and medical procedures) | 1 | 4
SHOULDER ARTHROPLASTY (Surgical and medical procedures) | 0 | 1
SPINAL FUSION SURGERY (Surgical and medical procedures) | 0 | 1
STERNOTOMY (Surgical and medical procedures) | 0 | 1
TOE AMPUTATION (Surgical and medical procedures) | 2 | 0
TRANSURETHRAL PROSTATECTOMY (Surgical and medical procedures) | 1 | 0
VASCULAR STENT INSERTION (Surgical and medical procedures) | 1 | 0
AIR EMBOLISM (Vascular disorders) | 0 | 1
AORTIC STENOSIS (Vascular disorders) | 3 | 3
ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 1
ARTERIAL THROMBOSIS LIMB (Vascular disorders) | 0 | 1
ARTERIOSCLEROSIS (Vascular disorders) | 1 | 1
ARTERIOVENOUS FISTULA (Vascular disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 1
FEMORAL ARTERY OCCLUSION (Vascular disorders) | 0 | 1
HAEMATOMA (Vascular disorders) | 5 | 1
HAEMORRHAGE (Vascular disorders) | 1 | 2
HYPERTENSION (Vascular disorders) | 1 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 1 | 1
HYPOTENSION (Vascular disorders) | 5 | 3
INTERMITTENT CLAUDICATION (Vascular disorders) | 3 | 0
ISCHAEMIA (Vascular disorders) | 1 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 2 | 3
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 | 0
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 | 2
SHOCK HAEMORRHAGIC (Vascular disorders) | 0 | 1
THROMBOPHLEBITIS (Vascular disorders) | 1 | 1
THROMBOSIS (Vascular disorders) | 0 | 1
VASCULAR DISSECTION (Vascular disorders) | 14 | 11
VESSEL PERFORATION (Vascular disorders) | 8 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Coronary PCI Guided by OCT (N=1233) | Coronary PCI Guided by Angiography (N=1254)
CARDIAC ENZYMES INCREASED (Investigations) | 71 | 73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/77/NCT03507777/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT03507777/SAP_001.pdf